CLINICAL TRIAL: NCT00119249
Title: A Phase II Study of BAY 43-9006 (NSC 724772) in Unresectable Stage III and IV Melanoma (IND 69,869)
Brief Title: Sorafenib in Treating Patients With Stage III or Stage IV Melanoma That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02659; NYWCCC-NYU-0438; N01CM62204 (NIH); CDR0000434613 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Stage III Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — Sorafenib

ARMS (1):
- Treatment (sorafenib tosylate) (Experimental): Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. This phase II trial is studying how well sorafenib works in treating patients with stage III or stage IV melanoma that cannot be removed by surgery

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of sorafenib, in terms of anti-tumor effects and proportion of clinical responses, in patients with previously untreated unresectable stage III or stage IV melanoma.

SECONDARY OBJECTIVES:

I. Correlate the efficacy of this drug with the presence of mutant or wild-type BRAF gene in tumors of these patients.

II. Determine the toxicity profile of this drug in these patients. III. Correlate serum cryptic collagen epitopes with the extent of tumor burden, invasion, and metastasis in patients treated with this drug.

IV. Determine the potential of serum cryptic collagen epitopes to serve as a surrogate marker for monitoring the course of disease in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to presence of BRAF gene mutation in tumor sample (yes vs no).

Patients receive oral sorafenib twice daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed annually.

PROJECTED ACCRUAL: A total of 26-74 patients (13-37 per stratum) will be accrued for this study within 5.2-18.5 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed unresectable melanoma

  * Stage III or IV disease
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion > 20 mm by conventional techniques OR > 10 mm by spiral CT scan
* Disease amenable to biopsy (first 13 patients in each stratum only)
* Brain metastases allowed provided the following criteria are met:

  * Disease has remained radiologically stable for ≥ 6 weeks after completion of whole-brain radiotherapy and remains stable at the time of study entry
  * No mass effect present by radiology
  * No requirement for steroid therapy to control symptoms of brain metastases
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 3 months
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No evidence of bleeding diathesis
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 2 times ULN
* Creatinine ≤ 1.5 times ULN
* No uncontrolled hypertension
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness that would preclude study compliance
* No pre-existing non-hematological dysfunction ≥ grade 2
* No ongoing or active infection
* No history of serious allergic reaction to eggs
* Able to swallow pills
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or other non-invasive carcinoma
* No other uncontrolled illness
* Not specified
* No prior systemic chemotherapy for metastatic disease
* See Disease Characteristics
* See Disease Characteristics
* No other concurrent investigational agents
* No concurrent therapeutic anticoagulation
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) defined as is either a complete or a partial response using RECIST criteria | 56 days
  The overall response rate along with subgroup-specific response rates will be estimated at the end of the trial along with 95% confidence interval.

SECONDARY OUTCOMES:
Time to progression | From the first day of treatment until the first documentation of disease progression, assessed up to 3.5 years
  Kaplan-Meier estimates will be calculated for time to progression and overall survival, and medians, along with two-sided 95% confidence intervals, will be reported.
Toxicity assessed using NCI CTCAE version 3.0 | Up to 3.5 years
  All adverse events without regard to causal relationship and by causal relationship to study drugs will be summarized.
Changes in BRAF, P-MAPK, CDK4, and cyclin D1 levels | Baseline and up to 3.5 years
  The proportion of patients with decreases in levels of BRAF, CDK4, or phospho-MAPK will be estimated along with 95% confidence intervals.
Overall survival | Up to 3.5 years
  Kaplan-Meier estimates will be calculated for time to progression and overall survival, and medians, along with two-sided 95% confidence intervals, will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pavlick, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Ott PA, Hamilton A, Min C, Safarzadeh-Amiri S, Goldberg L, Yoon J, Yee H, Buckley M, Christos PJ, Wright JJ, Polsky D, Osman I, Liebes L, Pavlick AC. A phase II trial of sorafenib in metastatic melanoma with tissue correlates. PLoS One. 2010 Dec 29;5(12):e15588. doi: 10.1371/journal.pone.0015588. PMID 21206909